CLINICAL TRIAL: NCT05818020
Title: Fighting Cancer Resistance: Multidisciplinary Integrated Platform for a Technological Innvovative Approach to Oncotherapies
Brief Title: Multidisciplinary Integrated Platform for a Technological Innvovative Approach to Oncotherapies
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: Campania Oncoterapie; 40/19oss (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Biologic
Keywords: Realization of a regional "Technology platform"

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is multicentric, observational, and retro- prospective study.

DETAILED DESCRIPTION:
The project aims to develop a regional platform for innovative disease treatment oncology. In particular, an integrated platform will be created with several complementary skills among them, which have as their common objective to increase knowledge and the possibilities of surgery for certain types of cancer.

The actions implemented in this project will be as follows:

* Improvement of primary and secondary prevention strategies with precocious diagnostic devices;
* Optimization of therapeutic treatments by custom drawing of the scheme therapeutic;
* Improved therapeutic efficacy for high social impact resistant neoplasms development of innovative treatments such as personalized therapeutic vaccines and small molecules;
* Improving patient compliance and quality of life accompanied by less need of hospitalization of the patient himself with consequent decongestion of hospital admissions;
* Reduction of health costs as a result of early diagnosis and new therapies more effective and less invasive;
* Increasing regional health and technological attractiveness in a high bio-medical sector social and health impact.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any of the following diseases:

  1. breast cancer;
  2. melanoma;
  3. hepatocarcinoma;
  4. gynecological cancer;
  5. colorectal cancer;
  6. lung cancer.
  7. sarcoma;
  8. pancreatic tumor;
  9. tumor of endocrine glands (thyroid);
  10. digestive system tumor (classifying rare ones);
  11. urological and/or male genital tumor (classifying rare ones);
  12. female genital tumor (classifying rare ones);
  13. rare skin tumor;
* Signature of the informed consent for the study.
* Age 18 years
* Biological material leftover from biopsy or surgery, and the residual to the activities of clinical assistance analysis.
* No ongoing treatment for oncological diseases at the time of collection.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for the present study:

* Patients aged < 18 years;
* Patients who have not signed the informed consent;
* Positive history of previous neoplasms (only for "naive" patients);
* Positive history of synchronous/metachronous oncological pathologies different from those specified for recruitment (only for "naive" patients);
* Ongoing immunosuppressive therapy (only for "naive" patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in the study were diagnosed with a tumor pathology between the following: Breast cancers, melanomas (cutaneous and non-cutaneous), liver tumors, bile duct tumors, colorectal tumors, lung tumors, sarcomas, pancreatic tumors, tumors of the endocrine glands (thyroid), digestive system tumors (classifying rare ones), urological and male genital tumors (classifying rare ones), female genital tumors (classifying rare ones); rare skin tumors.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Sampling of biological material from cancer patients. | 3 years
  Sampling size and type of biomaterials, residues in diagnosis and/or clinical activities care, collected by cancer patients and properly stored will include:
  - cells and/or tissue fragments during surgical excision (with "open" approach/ laparoscopic/ robotic) of the tumor or parts of the same tissue
Sampling of biological material from cancer patients. | 3 years
  Sampling size and type of biomaterials, residues in diagnosis and/or clinical activities care, collected by cancer patients and properly stored will include:- blood, cell samples, urine/other biological liquids (saliva, excreted, ascites, pleural fluids, etc.) and faeces,
Sampling of biological material from cancer patients. | 3 years
  Sampling size and type of biomaterials, residues in diagnosis and/or clinical activities care, collected by cancer patients and properly stored will include:- samples fixed in formalin and included in paraffin (Formalin-fixed paraffin-embedded, FFPE).
Identification of biomarkers to be used for the development of early diagnostic systems | 3 years
  The alteration of the levels of biomarkers, measured by the use of analytical techniques based on mass spectrometry, and the correlation of such levels measured against control samples will allow the development and training of advanced statistics models to identify and define the type and the status of the oncological pathology.
Monitoring the progress of drug therapies | 3 years
  The identification of biomarkers used to monitor the drug therapie defined as "pharmacometabolomics" will allow to calibrate finely and optimize the selection of therapeutic protocols allowing to reduce the costs of prescription and assistance, while improving the patient's health.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Normanno, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (3):
- Italy (3):
  - Clinica Padre Pio srl, Mondragone, CE
  - Pineta Grande Hospital, Castel Volturno, Napoli
  - Istituto Nazionale Tumori | "Fondazione Pascale", Napoli